CLINICAL TRIAL: NCT06550245
Title: The Malleability of Social Group Understanding in Infancy and Early Childhood
Brief Title: Babies' Brain Responses to Strangers
Status: Recruiting | Type: Observational
Sponsor: University of California Santa Cruz (Other)
Responsible Party: Sponsor
Other Study IDs: HS-FY2023-23 Study 2
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Infant Development

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Infants observing familiar and unfamiliar racial groups — All infants will see videos of people from familiar and unfamiliar racial backgrounds. Depending on the caregiver's race, infants will be assigned to see people who are from the same racial background as their caregiver (i.e., familiar) and people who are not.

SUMMARY:
Researchers at the Diversity in Development Lab at UC Santa Cruz are investigating how babies' brain activities respond to people from familiar and unfamiliar racial backgrounds.

DETAILED DESCRIPTION:
The goal of this observational study is to learn how infants' brain activities, as captured by EEG, differ for familiar or unfamiliar racial group in typically developing infants. The main questions of the study are:

* Will infants show greater event-related desynchronization (i.e., more motor system activation), frontal theta synchronization (i.e., more attention), and more positive frontal alpha asymmetry (i.e., more approach motivation) to familiar than unfamiliar racial group?
* How does infants' exposure to racial diversity in their social network and neighborhoods relate to these EEG activities? Participants will visit a laboratory at the UC Santa Cruz campus for this study. Infants will put an EEG cap on and watch about 15 minutes of videos, in which people from different racial backgrounds do different actions (e.g., grabbing an object, saying hi and approaching closer, and playing peek-a-boo). Caregivers will be asked to fill out a demographic form and a social network survey.

ELIGIBILITY:
Inclusion Criteria:

* typically developing
* age 7 to 12 months
* at least 37 weeks gestation

Exclusion Criteria:

* any known developmental delays
* less than 37 weeks gestation

Ages: 7 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: community sample from the larger Santa Cruz area
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mu event related desynchronization | Through study completion, an average of 10 years.
  EEG oscillation in alpha power over central regions
Frontal theta synchronization | Through study completion, an average of 10 years.
  EEG oscillation in theta power over frontal regions
Frontal alpha asymmetry | Through study completion, an average of 10 years.
  left and right hemispheric difference in EEG oscillation in alpha power in the frontal regions

CONTACTS AND LOCATIONS:
Overall Officials: Hyesung Hwang, PhD, Principal Investigator — University of California Santa Cruz
Locations (1):
- Social Science 2 Building, Santa Cruz, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that are anonymized and underlie results in a publication will be shared through open science framework (OSF)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available within a period of 10 years. Anonymized aggregate data will be available indefinitely. No identifiable data will be shared.
Access Criteria: All anonymized data will be available once study has been published and will be available indefinitely.

REFERENCES:
- [Background] Hwang HG, Debnath R, Meyer M, Salo VC, Fox NA, Woodward A. Neighborhood racial demographics predict infants' neural responses to people of different races. Dev Sci. 2021 Jul;24(4):e13070. doi: 10.1111/desc.13070. Epub 2020 Dec 16. PMID 33277794